CLINICAL TRIAL: NCT04600271
Title: Risk Factors of Acute Kidney Injury After Major Elective Non-Cardiac Surgery : A Prospective Observational Study
Brief Title: Acute Renal Injury After Major Elective Non-Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dilan Büyük, Resident at Anesthesiology and Reanimation, Istanbul University
Other Study IDs: 2019/747
Record Dates: First submitted 2020-10-11; First posted 2020-10-23 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Acute Renal Injury
Keywords: colloids; mean arterial blood pressure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Crystalloid Solutions; Diuretics; Norepinephrine; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients over the age of 18 and who undergone major elective non-cardiac abdominal surgery.
  Interventions: Drug: Crystalloid Solutions; Drug: Colloid Blood Volume Expanders; Other: blood replacement; Drug: Diuretic; Drug: noradrenaline; Drug: Non-Steroidal Anti-Inflammatory Analgesics

INTERVENTIONS:
Drug: Crystalloid Solutions — exposure
Drug: Colloid Blood Volume Expanders — exposure
Other: blood replacement — exposure
Drug: Diuretic — exposure
Drug: noradrenaline — exposure
Drug: Non-Steroidal Anti-Inflammatory Analgesics — exposure

SUMMARY:
The study is planned to be a single-center study and includes patients who underwent major surgery within Istanbul University Istanbul Faculty of Medicine with an invasive arterial line. Our aim to define the incidence of acute renal injury in our setting and to investigate the risk factors listed in detailed description. After obtaining written informed consent from the patients, preoperative risk factors will be notes. Following standard anesthesia monitoring as well as routine anesthesia induction and maintenance, invasive arterial monitoring will be performed due to the major surgery and hemodynamic values will be recorded throughout the surgery. The primary outcome will be acute renal injury based on KDIGO's (Kidney Disease: Improving Global Outcomes) definition of acute renal damage. Postoperative data regarding this outcome as well as additional data listed in detailed description will be collected.

DETAILED DESCRIPTION:
The study is a single-center study that observes patients who undergo major abdominal surgery within Istanbul University Istanbul Faculty of Medicine.

Standard anesthesia monitoring (NIBP, SPO2(oxygen saturation by pulse oximetry), ECG) will be applied to the patients taken to the operation room. Routine anesthesia induction and maintenance will be performed by the anesthetist responsible for the patients. After anesthesia induction, invasive arterial monitoring will be performed.

Our data collection and recording will be as follows: preoperative, intraoperative, postoperative.

In the preoperative section;

* Age, gender, height, weight, BMI of the patient
* ASA (American Society of Anesthesiologists) classification, additional diseases and functional capacity
* Drugs used (ACE-İ, ARB (angiotensin receptor blocker), Statin, B-blocker, NSAID)
* Entry creatinine and eGFR (estimated glomerular filtration rate) calculated with CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration)
* Entry hemoglobin, lymphocyte, CRP (C reactive protein)
* The presence of ascites in the abdomen

In the intraoperative section;

* Surgery (gynecological oncology surgery, gastrointestinal surgery, genitourinary surgery) and its duration
* Applied form of anesthesia (general-regional)
* Liquids given during the operation (Crystalloid (isotonic, isolyte, lactated ringer), colloid, albumin) and their amounts oNoradrenaline requirement
* Use of diuretic, NSAID
* Blood transfusion
* Total amount of bleeding during the operation
* First arterial blood gas electrolytes taken due to routine major surgery
* The lowest amount of hemoglobin seen during the operation
* Routine invasive artery monitorization due to major surgery, and mean arterial pressure In the postoperative section;
* Requirement of intensive care
* Blood transfusion requirement
* Noradrenaline requirement
* Use of diuretic and NSAID
* Electrolyte values in the first blood gas taken routinely
* Creatinine value immediately after the surgery and at 24th and 48th hours
* First 48-hour urine output The diagnosis of acute renal injury is based on KDIGO's definition of acute renal damage. By analyzing from this information, significant risk factors for acute renal damage are identified and measures are taken against them.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years
* Patients who are ASA I-III
* Patients who have undergone major noncardiac surgery
* Patients who need post-operative intensive care follow-up due to major surgery or long surgery
* Patients diagnosed with CKD but do not need routine hemodialysis

Exclusion Criteria:

* Age of <18 years
* Patients who have undergone minor surgery
* Surgeries which lasts <30 minutes
* Patients who will be hospitalized less than two days postoperatively
* Patients who need routine hemodialysis due to CKD
* Patients who had renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone non-cardiac major surgery in Istanbul University Faculty of Medicine will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Acute renal injury | 48 hours
  Acute renal injury description will be made with KDIGO criteria.

SECONDARY OUTCOMES:
Hospital stay | 30-90 days
  Will be noted as days.
ICU stay | 30-90 days
  Will be noted as days.
Chronic Kidney Disease | up to 1 year
  will be noted after postoperative period.
Mortality | 30-90 days
  will be noted in the hospital period.
Complication after surgery | 30-90 days
  will be noted in the hospital period.

CONTACTS AND LOCATIONS:
Overall Officials: Mukadder Orhun Sungur, Assos. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine Departmant of Anesthesiology and Reanimation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hobson C, Ruchi R, Bihorac A. Perioperative Acute Kidney Injury: Risk Factors and Predictive Strategies. Crit Care Clin. 2017 Apr;33(2):379-396. doi: 10.1016/j.ccc.2016.12.008. PMID 28284301
- [Background] Goren O, Matot I. Perioperative acute kidney injury. Br J Anaesth. 2015 Dec;115 Suppl 2:ii3-14. doi: 10.1093/bja/aev380. PMID 26658199
- [Result] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335